CLINICAL TRIAL: NCT03046225
Title: Acute Effects of Transcutaneous Electric Nerve Stimulation in Patients Rehabilitation After Total Knee Arthroplasty.
Brief Title: Transcutaneous Electrical Nerve Stimulation After Total Knee Arthroplasty.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-0104
Record Dates: First submitted 2016-11-29; First posted 2017-02-08 (Estimated); Results first posted 2018-03-22 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2017-02

CONDITIONS: Transcutaneous Electric Nerve Stimulation; Pain
MeSH Terms: conditions — Pain | interventions — Transcutaneous Electric Nerve Stimulation; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electrical stimulation (Experimental): This group received application of transcutaneous electrical nerve stimulation (TENS) associated with conventional physical therapy (continuous passive movement device and exercises).
  Interventions: Device: Transcutaneous electrical nerve stimulation; Device: Continuous passive movement device; Other: Exercises
- Physical therapy (Active Comparator): This group received only conventional physical therapy (continuous passive movement device and exercises).
  Interventions: Device: Continuous passive movement device; Other: Exercises

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation — TENS was applied in the conventional mode, through two self-adhesive electrodes of size 5x9cm positioned parallel to the lumbar spine, on the nerve roots of L3, L4 and L5, with frequency of 100 Hz and pulse duration of 100 μs, for 30 minutes. The intensity was adjusted according to the maximum tolerance of the patient and was gradually increased, with his permission, during the application time.
  Other Names: TENS
  Arms: Electrical stimulation
Device: Continuous passive movement device — CPM device was used for 30 minutes and realized continuous passive flexion and extension of the operated knee.
  Other Names: CPM
Other: Exercises — Active exercises of plantar flexion and dorsal flexion of the ankles, adduction and abduction of the hips and flexion and extension of the operated knees. All exercises were performed in 10 repetitions, with the patient positioned in the supine position in the bed.

SUMMARY:
Total knee arthroplasty (TKA) consists of a surgical replacement of this joint by a prosthesis, and it is mainly carried out in cases of knee osteoarthrosis. In the postoperative period of TKA, the pain is intense and limits the mobility of patients, so the analgesia is one of the goals of the physical therapy. One of the alternatives available for pain management is the transcutaneous electrical nerve stimulation (TENS), characterized by the application of an electric pulsed current through electrodes positioned on the skin. Therefore, the present study aims to evaluate the acute effects of TENS associated with conventional physical therapy compared with conventional physical therapy on the pain level, knee range of motion and administration of morphine in the rehabilitation of patients after TKA.

DETAILED DESCRIPTION:
The study included patients who underwent TKA surgery in the Hospital de Clínicas de Porto Alegre (HCPA) and met the study eligibility criteria. The sample was randomly divided into experimental group, which received conventional physical therapy associated with the application of TENS, and control group, which held only conventional physical therapy, both on the first day after the surgery. The pain level, the range of motion of the operated knee and the Administration of morphine.

The experimental group received TENS application held by two self-adhesive electrodes size 5x9cm positioned parallel to the lumbar spine, on the nerve roots L3, L4 and L5. TENS was applied in conventional mode, emitting a pulsed biphasic, symmetrical rectangular wave with frequency of 100 Hz and pulse duration of 100 µs, for 30 minutes. The intensity was set according to the tolerance of the patient and was gradually increased during the application. The device used was the Neurodyn II model, by Ibramed.

Subsequently, the conventional physical therapy was performed, with the use of the CPM device and performing exercises. The CPM device was used for 30 minutes, and realized continuous passive flexion and extension of the operated knee. The amplitudes of these movements were gradually increased in accordance with the tolerance of the patient. The device used was Spectra model, by Kinetec.

Then, the patients realized active exercises of plantar flexion and dorsal flexion of the ankles and adduction and abduction of the hips, isometric exercises of flexion and extension of the operated knee and active exercises of flexion and extension of the non-operated knee. All exercises were performed in 10 repetitions, with the patient positioned in the supine position in the bed.

The control group received only conventional therapy consisting of the use of the CPM device in the operated leg and the exercises in both lower limbs, identical to those performed in the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent TKA surgery due to primary or secondary gonarthrosis; Both sexes; Age between 40 and 90 years.

Exclusion Criteria:

* Patients who refused to participate of the study; Indication of TKA for fractures and bone tumors; TKA review surgery; Infection during the postoperative period; Congenital anatomical alterations; Neurological disorders; Lack of understanding of commands; Sensitivity alterations in the lumbar spine or lower limbs; Decompensated heart disease or cardiac pacemaker use.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-05; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was carried out at the Hospital de Clínicas de Porto Alegre Hospital (HCPA), Rio Grande do Sul, Brazil. Evaluations and interventions occurred between May and September 2016.
Period: Overall Study
Arm/Group | Electrical Stimulation | Physical Therapy
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Electrical Stimulation | Physical Therapy | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.8 (7.4) | 66.5 (7.4) | 67.1 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 3 | 0 | 3
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 30.7 (3.7) | 32 (4.3) | 31.3 (4)
Femoral nerve block [Count of Participants; unit: Participants] | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Level From Baseline to 90 Minutes
Description: It was measured by Visual Analogue Pain Scale (VAS), which has scores ranging from zero (which means "no pain") to 10 (which means "worst possible pain"). Two evaluations of the pain level were performed in each group, before and after the interventions.
Time Frame: 90 minutes
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Electrical Stimulation | Physical Therapy
Number analyzed (Participants) | 13 | 13
Units on a scale | 3.1 (2.6) | 3.3 (2.7)

2. Secondary Outcome: Number of Participants Who Received Morphine Within 24 Hours
Description: It was evaluated based on the information found in patients' electronic records, considering whether they received morphine during the 24 hours following the interventions or not.
Time Frame: 24 hours
Measure: Number; unit: Participants
Arm/Group | Electrical Stimulation | Physical Therapy
Number analyzed (Participants) | 13 | 13
Participants | 6 | 8

3. Secondary Outcome: Change in Knee Range of Motion From Baseline to 30 Minutes
Description: It was extracted from the continuous passive movement device display. During the use of the continuous passive movement device (CPM), from the observation of the digital display in its control, the degrees of amplitude reached in the passive movements of flexion and extension of the knee submitted to the surgery were extracted.
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Electrical Stimulation | Physical Therapy
Number analyzed (Participants) | 13 | 13
Degrees | 46.2 (10.4) | 44.9 (6.2)

ADVERSE EVENTS:
Time Frame: 24 hours.
Description: The exclusion criteria of the experiment included contraindications for the use of TENS: neurological disorders; lack of understanding of commands; sensitivity alterations in the lower limbs; decompensated heart disease or cardiac pacemaker use. None of the included subjects presented those conditions, therefore the risk of adverse events was zero, since they were exposed to no risk therapies and were followed by a therapist during the data collection.
Arm/Group | Electrical Stimulation | Physical Therapy
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

LIMITATIONS AND CAVEATS:
The subjects had difficulty to understand Visual Analogue Pain Scale, the sample was small, and there was not a TENS placebo group, which could allow other comparisons on the effectiveness of TENS in this population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes